CLINICAL TRIAL: NCT01855841
Title: Prevention of Post-ERCP Acute Pancreatitis by Heme-oxygenase Activation Through the Administration of Hemin : a Prospective, Randomized Double Blind Controlled Trial
Brief Title: Hemin to Prevent Post-ERCP (Endoscopic Retrograde Cholangiopancreatography) Acute Pancreatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Lemmers Arnaud, MD, PhD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hemin_AP
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: ERCP; virgin papilla; risk of post-ERCP acute pancreatitis
MeSH Terms: interventions — Hemin; Heme; heme arginate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemin (Active Comparator): A peripheral perfusion of 4mg/kg of hemin (Normosang) diluted in 100mL NaCL (sodium chloride) 0.9% will be administered in 30-60minutes as soon as possible after the end of the ERCP, followed by 100mL of NacL 0.9% to flush the vein
  Interventions: Drug: Hemin
- Placebo (Placebo Comparator): The same amount of NaCl 0.9% (100 ML followed by a flushing perfusion of 100mL) will be perfused to the patient as soon as possible after the end of the ERCP
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Hemin — A single perfusion of 4mg/kg hemin diluted in 100mL of NaCl 0.9% administered as soon as possible after the end of the ERCP followed by 100mL of NaCL 0.9% to flush the vein
  Other Names: Haemin; Normosang
  Arms: Hemin
Drug: placebo — A single perfusion of 100mL of NaCl 0.9% administered as soon as possible after the end of the ERCP followed by 100mL of NaCL 0.9% to flush the vein
  Other Names: saline
  Arms: Placebo

SUMMARY:
ERCP (endoscopic retrograde cholangiopancreatography) has been largely demonstrated to be effective in multiple bilio-pancreatic indications. However, one of the feared complication of this technique is acute pancreatitis, which happens in 5 to 25% of cases. Some patient groups have been demonstrated to present a higher risk linked to individual factors or to the procedure. Some interventions (endoscopic or pharmacologic) have been evaluated to reduce the incidence of this complication but each has his own inconvenient. Recently, the activation of heme oxygenase (HO) by intraperitoneal administration of hemin has been demonstrated to be effective in prevention and treatment of acute pancreatitis mice models. This protective effect has been associated to intrapancreatic HO-1 positive macrophage recruitment activated by hemin. The investigators thus propose to conduct a prospective randomized double blind controlled trial to demonstrate a protective effect of hemin administration against post-ERCP acute pancreatitis in high risk patients.

DETAILED DESCRIPTION:
Patients for who a pancreatic stent placement is indicated will be excluded from the study.

The aims of this study are: 1) to study in a pathophysiologic point of view the activation of HO-1 by hemin in human and its protective effect in post-ERCP acute pancreatitis incidence. 2) to use the human situation of post-ERCP acute pancreatitis as early pancreatitis model to study the administration of hemin as treatment of acute pancreatitis in general.

ELIGIBILITY:
Inclusion Criteria: one or more factors of >10% post-ERCP acute pancreatitis risk:

* former episode of acute pancreatitis
* former episode of post-ERCP acute pancreatitis
* normal bilirubin level
* main pancreatic duct injection
* endoscopic biliary sphincteroplasty (balloon dilation of biliary sphincter)
* precut papillotomy
* pancreatic sphincterotomy

Exclusion Criteria:

* patient for whom a pancreatic stent is inserted (Sphincter of Oddi dysfunction, ampullectomy)
* ongoing acute pancreatitis
* chronic pancreatitis (Cremer classification >=2)
* age < 18 y/o
* pregnancy
* hemin allergy
* severe renal failure (MDRD<30ml/min/1.73m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Incidence of post-ERCP acute pancreatitis | at day 1 post-ERCP
  Post-ERCP acute pancreatitis is defined by an abdominal pain compatible with pancreatitis and the elevation of seric lipases more than 3 times the upper limit of normal on days 1 post-ERCP.

SECONDARY OUTCOMES:
severity of post-ERCP acute pancreatitis | during the hospital stay (up to 2 months)
  If post-ERCP acute pancreatitis happens, all parameters of severity will be recorded (clinical, biological, intra-abdominal collections seen on abdominal scanner/magnetic resonance, organ failure, need for ICU hospitalization, need for further treatment: surgery/endoscopy/radiological drainage?)
length of stay | during the hospitalization (up to 2 months)
  the length of stay in the hospital will be recorded. if a complication occurs (post-ERCP acute pancreatitis or other, it will be recorded)
safety of hemin administration | within 7 days
  Few side effects of hemin are known (headache, superficial thrombophlebitis in the perfused vein); they will be recorded as well as other unexplained clinico-biological events

OTHER OUTCOMES:
number of patients with post-ERCP acute pancreatitis and adverse event at interim analysis | after 100 patients
  After having randomized 50 patients by arm, an interim analysis will be conducted to evaluate the safety (superficial venous thrombophlebitis, headache, unexpected adverse events)and need to complete the study (depending on the results on post-ERCP acute pancreatitis incidence)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Lemmers, MD,PhD, Principal Investigator — Erasme Hospital, Université libre de Bruxelles (ULB), Brussels, Belgium; Jacques Devière, MD, PhD, Study Chair — Erasme Hospital, Université Libre de Bruxelles (ULB), Brussels, Blegium
Locations (6):
- Belgium (5):
  - CHU Brugmann, Brussels
  - Erasme Hospital, Université Libre de Bruxelles (ULB), Brussels
  - Centre Hospitalier de Jolimont-Lobbes, Haine-St-Paul
  - Hôpital Ambroise Paré, Mons
  - ISPPC CHU Vésale, Montigny-le-Tilleul
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yared RA, Chen CC, Vandorpe A, Arvanitakis M, Delhaye M, Viesca MFY, Huberty V, Blero D, Toussaint E, Hittelet A, Verset D, Margos W, Le Moine O, Njimi H, Liao WC, Deviere J, Lemmers A. Intravenous Hemin, a potential heme oxygenase-1 activator, does not protect from post-ERCP acute pancreatitis in humans: Results of a randomized multicentric multinational placebo-controlled trial. Pancreatology. 2024 May;24(3):363-369. doi: 10.1016/j.pan.2024.02.009. Epub 2024 Feb 15. PMID 38431445